CLINICAL TRIAL: NCT03533140
Title: Low Level Transcutaneous Electrical Vagus Nerve Stimulation To Suppress Atrial Fibrillation
Brief Title: Postoperative Atrial Fibrillation Suppression By Nerve Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alfred A Kocher, MD, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1 KlinPruefplanProtocol6
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DUCEST Neurostimulator V Group A (Active Comparator)
  Interventions: Device: DUCEST Neurostimulator V Group A
- DUCEST Neurostimulator V Group B (Sham Comparator)
  Interventions: Device: DUCEST Neurostimulator V Group B

INTERVENTIONS:
Device: DUCEST Neurostimulator V Group A — The DUCEST Neurostimulator V needle-electrodes are applied post-operatively to stimulate the R.auricularis of the vagus nerve located at the Fossa triangularis. Connecting the needle-electrode cables to the Neurostimulator V activates the device. (The stimulation intensity can be adjusted from 0,05mA to 1,2mA, default value is 0,4mA). The starting stimulation intensity will be adjusted to 1mA and takes place at 1Hz continuously for 40 minutes, followed by a 20 minute break. The built-in 3V battery lasts for approx. 14 days. After 7 days the electrodes are replaced and applied to the other ear of the patient. A plaster with a plastic mounting clip is attached on the shoulder of the patient. The Neurostimulator is connected to the mounting clip. After 14 days or at hospital discharge of the patient, the device is unmounted and the needle-electrodes are removed.
  Arms: DUCEST Neurostimulator V Group A
Device: DUCEST Neurostimulator V Group B — The DUCEST Neurostimulator V needle-electrodes are applied post-operatively at the Fossa triangularis. Connecting the needle-electrode cables to the Neurostimulator V activates only the signal lamp but not the device.
  Arms: DUCEST Neurostimulator V Group B

SUMMARY:
The current study will evaluate the potential of stimulating the R.auricularis of the vagus nerve located at the Fossa triangularis to ameliorate or suppress AF in the study Population!

DETAILED DESCRIPTION:
Scientific Background Nearly 30% of patients undergoing coronary artery bypass grafting (CABG), 40% of patients undergoing valvular heart surgery and over 50% of patients with combined coronary and valvular procedures develop atrial fibrillation (AF).

Postoperative AF occurs mostly due to conditions like chronic kidney diseases, emergency surgery, age >75 years, cardiopulmonary bypass time >180 min and due to lacking postoperative application of aldosterone- and beta-blockers.

An overview of pre- intra- and postoperative risks for AF is listed in

Table 1: Pre-, intra-, postoperative risks for AF.

Preoperative High age Male gender Previous cardiac surgery Valvular heart disease Chronic lung disease Chronic renal failure Leſt atrium enlargement Leſt ventricular hypertrophy Withdrawal of beta-blocker medication History of AF Hypertension Obesity Diabetes Metabolic Syndrome

Intraoperative Endotracheal tube insertion Intraoperative IABP Leſt ventricular venting Aortic cross-clamp time Extracorporeal circulation Myocardial ischemia Venous cannulation Damage to the atrium Excess inotropic requirements Acute volume change

Postoperative Return to intensive care unit Ventilation longer than 24 hours Volume overload Pneumonia Electrolyte imbalances Imbalance of auton. nervous system Atrial extrasystole Increased postop adrenergic status Increased aſterload Inflammation Hypotension

Several theories describe the emergence of AF like "multiple-wavelet re-entry", "focal mechanism" and "mother rotor" but the exact underlying mechanisms are still not well understood.

Prevention and treatment of postoperative AF are managed with conservative medication therapies including e.g. beta-blockers and other clinical interventions include radio frequency catheter ablation, cardioversion and occlusion of the left atrial appendage.

A novel approach for suppression of AF utilizing low-level transcutaneous electrical vagus nerve stimulation has been described recently in the Journal of the American College of Cardiology. The newly developed "DUCEST Neurostimulator V" device (manufactured by Biegler Medizinelektronik GmbH Mauerbach, Austria) offers similar action as in. This Neurostimulator device is designed to emit small direct current electrical pulses (0-1,2mA) to stimulate the R.auricularis of the vagus nerve located at the Fossa triangularis. The target population are patients with de-novo postoperative AF. The stimulation is achieved with the attachment of two needle- electrodes and connection of the electrodes to the Neurostimulator.

Following the stimulation of the vagus nerve positive effects were already achieved in chronical wound healing, peripheral artery occlusive disease (PAOD), Claudicatio intermittens (CI) and chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* De-novo postoperative AF
* CABG or aortic valve replacement
* Age of 18-80 years
* Willing and able to understand, sign and date the informed consent form that has been approved by the institutional review board

Exclusion Criteria:

* Pacemaker or ICD
* Impaired EF < 30%
* Patients with acute myocardial infarction within the past 14 days
* Pregnant or lactating patients
* Any condition that, in the judgement of the investigator, would place the patient at undue risk
* Any concurrent disease or condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the study
* Treatment and/or an uncompleted follow-up treatment of any investigational therapy within 6 months before procedure and intent to participate in any other investigational drug or cell therapy study during the follow-up period of this study
* Active participation in other Research therapy for cardiovascular repair/regeneration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Atrial Fibrillation events in routine ECG and continous HOLTER ECG for the length of the hospital stay. | 07-14 days post operative
  Patients are randomized to a treatment or a sham group. The corresponding device is prepared by a third person according to the double-blind setting for the surgeon. The DUCEST Neurostimulator V needle-electrodes are applied post-operatively to stimulate the R.auricularis of the vagus nerve located at the Fossa triangularis. Connecting the needle-electrode cables to the Neurostimulator V activates the device. (The stimulation intensity can be adjusted from 0,05mA to 1,2mA, default value is 0,4mA). The starting stimulation intensity will be adjusted to 1mA and takes place at 1Hz continuously for 40 minutes, followed by a 20 minute break. After 7 days the electrodes are replaced and applied to the other ear of the patient. A plaster with a plastic mounting clip is attached on the shoulder of the patient. The Neurostimulator is connected to the mounting clip. After 14 days or at hospital discharge of the patient, the device is unmounted and the needle-electrodes are removed.

SECONDARY OUTCOMES:
Measurement of postoperative inflammation markes, using plasma values of CRP, TNF-alpha, IL-6, and IL-10 | 07-14 days post operative
  Inflammation markers will be assessed via laboratory blood sample testing at day 0 (at device attachment), +2 and +7 days post device attachment. CRP, TNF-alpha, IL-6, and IL-10 will be will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Kocher, MD, Principal Investigator — Surgeon

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03533140/Prot_000.pdf